CLINICAL TRIAL: NCT00407940
Title: ATHERO: Advanced Technology Halting Early Re-Stenosis and Occlusion. A Prospective Randomized Trial Comparing Silverhawk™ Atherectomy to CryoPlasty® Therapy for Lower Extremity Claudication
Brief Title: ATHERO: Advanced Technology Halting Early Re-Stenosis and Occlusion
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 007A
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Arterial Occlusive Disease; Intermittent Claudication
Keywords: Thrombosis; Claudication
MeSH Terms: conditions — Arterial Occlusive Diseases; Intermittent Claudication; Thrombosis | interventions — Angioplasty

INTERVENTIONS:
Device: Lower extremity Atherectomy and Cryoplasty

SUMMARY:
The rise of minimal access surgery has heralded the approval of a number of endovascular devices with similar indications. This is particularly true for the treatment of lower extremity ischemia. Comparable devices are selected for patient use somewhat arbitrarily, often dependent on industry influence. An unmet need is NON-industry sponsored prospective trials COMPARING devices head-to-head so that endovascular surgeons can even contemplate evidence-based device selection. At present, we seek to compare two new high-technology devices that are indicated to treat lower extremity arterial stenoses associated with claudication.

DETAILED DESCRIPTION:
Peripheral arterial disease affects more than 12 million Americans, and its incidence is growing annually. The male/female ratio of patients with claudication is just under 2/1. The arteries involved by atherosclerosis involve the arteries to the thigh and leg. These include the femoral and popliteal arteries. Fifty percent of people with femoral-popliteal PVD are symptomatic. Symptoms are typically related to exertional fatigue of thigh and calf muscles. These symptoms, referred to as claudication, seldom represent a life or even limb-threatening process. They do, however, result in significantly decreased productivity and an often devastating quality of life.

Traditional interventions for lower extremity claudication include technologies invented in the first half of the 20th century including surgical bypass; and those invented in the second half of the twentieth century, including balloon angioplasty and stenting. These interventions have substantial shortcomings. It is, however, relevant to note that endovascular (aka endoluminal or endovascular surgery) is becoming increasingly popular and gaining wide-spread support from vascular interventionalist societies wordwide.

The main shortcomings of angioplasty and stenting is the resultant inflammatory response. The mechanical injury to blood vessels is followed by a complex repair response comprising intimal vascular smooth muscle cell (VSMC) hyperplasia, vessel wall scarring and shrinkage of the vascular lumen, often resulting in reduced blood flow and subsequent muscle (or end organ) ischemia. Rodent, rabbit and large animal models have provided valuable insights into the pathophysiology of these responses.

The devices utilized in this protocol are both FDA approved for the procedures described in the protocol. The devices include the Silverhawk™ System (FoxHollow Technologies, Redwood City, CA) and the PolarCath™ Peripheral Dilatation System, Boston Scientific, Natick, Massachusetts). Hereafter both products will be referred to as the "Devices."

ELIGIBILITY:
Inclusion Criteria:

* The subject must give written informed consent and possess decision making capacity free of sedative or hypnotic agents.
* Age 18 years or older
* Candidate for angiography with intent-to-treat as determined by the Principle Investigator
* On angiography, ipsilateral to a symptomatic limb, a stenotic or occluded de novo or restenotic lesion in the common femoral artery, superficial femoral artery or above the knee popliteal artery measuring no longer than 10 cm (the upper limit of treatment in Cryoplasty pre-marketing)
* On angiography Lesion stenoses between 50% and 100% (inclusive)
* At least one runoff vessel
* Available for follow-up assessments

Exclusion Criteria:

* Contraindication to systemic anticoagulation e.g. history of documented hemorrhage requiring treatment within the past 30 days; history of a hereditary bleeding disorder or known bleeding diathesis; major surgery or trauma, open chest massage, ocular surgery or hemorrhagic retinopathy within the past 30 days; puncture at a non-compressible site within 48 hours prior to planned procedure; history of stroke, intracranial hemorrhage, or central nervous system structural abnormalities within the past 3 months
* History of endovascular surgery procedure or open vascular surgery on the index limb within the last 30 days
* History of significant acute or chronic kidney disease that would preclude contrast angiography
* Known allergy to contrast agents
* History of heparin-induced thrombocytopenia (HIT)
* Participation in any study of an investigational device, medication, biologic, or other agent within 30 days prior to randomization
* Any thrombolytic therapy within 30 days of randomization
* Pregnancy, lactation, or possession of any child bearing potential without evidence of surgical infertility or passage of 12 months since the last day of the subject's last menstrual period.
* Target lesion involving a dacron prosthesis or a prosthetic of unknown material
* Target lesion extending into the orifice of the profunda femoris artery
* Prisoner status
* Any other subject feature that in the opinion of the investigator should preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Primary target patency at 12 months. The "target" is the index stenotic lesion(s). Primary patency is defined as <50% residual stenosis by duplex (color-flow Doppler) scan analysis, with antegrade flow to the target vessel.

SECONDARY OUTCOMES:
Ankle Brachial Index (ABI) improvement by ≥0.15 at 3, 6 and 12 months compared to baseline
Change in Walking Impairment Questionnaire (WIQ) functional status scores from baseline at 3, 6 and 12 months
Complications: defined as adverse events (AEs) or serious adverse events (SAEs). Complications may or may not be device related
Cost to patient and hospital: Including operating room times and duration of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Niren Angle, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Medical Center, Hillcrest, San Diego, California, United States

REFERENCES:
- [Background] Laird J, Jaff MR, Biamino G, McNamara T, Scheinert D, Zetterlund P, Moen E, Joye JD. Cryoplasty for the treatment of femoropopliteal arterial disease: results of a prospective, multicenter registry. J Vasc Interv Radiol. 2005 Aug;16(8):1067-73. doi: 10.1097/01.RVI.0000167866.86201.4E. PMID 16105918
- [Background] Zeller T, Rastan A, Schwarzwalder U, Frank U, Burgelin K, Amantea P, Muller C, Flugel PC, Neumann FJ. Percutaneous peripheral atherectomy of femoropopliteal stenoses using a new-generation device: six-month results from a single-center experience. J Endovasc Ther. 2004 Dec;11(6):676-85. doi: 10.1583/04-1316R.1. PMID 15615558
- [Background] Muradin GS, Bosch JL, Stijnen T, Hunink MG. Balloon dilation and stent implantation for treatment of femoropopliteal arterial disease: meta-analysis. Radiology. 2001 Oct;221(1):137-45. doi: 10.1148/radiol.2211010039. PMID 11568332